CLINICAL TRIAL: NCT00283335
Title: CSP #363 - The VA HDL Intervention Trial (HIT): Secondary Prevention of Coronary Heart Disease in Men With Low HDL-Cholesterol and Desirable LDL-Cholesterol
Brief Title: The VA HDL Intervention Trial (HIT): Secondary Prevention of Coronary Heart Disease in Men With Low HDL-Cholesterol and Desirable LDL-Cholesterol
Acronym: HIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Parke-Davis (Industry); Fournier Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 363
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Gemfibrozil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemfibrozil (Active Comparator): 1200 mg slow-release gemfibrozil (Lopid-SR) once per day
  Interventions: Drug: gemfibrozil
- Placebo (Placebo Comparator): Matching placebo tablets taken once per day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: gemfibrozil
  Arms: Gemfibrozil
Other: Placebo — Matching placebo tablets taken once per day
  Arms: Placebo

SUMMARY:
This was a double-blind randomized trial comparing 1200 mg per day of gemfibrozil with placebo in 2531 men with coronary heart disease, an HDL-C of 40mg/dl or less, an LDL-C of 140 mg/dl or less, and triglycerides of 300mg/dl or less. The primary outcome was nonfatal myocardial infarction(MI) or death from coronary causes. The median follow-up was 5.1 years. There was a risk reduction of 22% in the primary outcome (p=.0006) and 24% risk reduction in the combined endpoint of stroke, MI, and CHD death. The rate of events was reduced by raising HDL-C and lowering triglycerides without lowering LDL-C (N Engl J Med 1999;341:410-418).

DETAILED DESCRIPTION:
Primary Hypothesis:

To determine if drug treatment aimed at raising HDL-cholesterol and lowering triglycerides will reduce the rate of heart attack and death in veterans with coronary heart disease (CHD) and a specific lipid profile characterized by normal levels of LDL-cholesterol and low levels of HDL-cholesterol.

Secondary Hypotheses:

To determine the effect of treatment on total mortality, unstable angina, CABG, PTCA, strokes and PVD, and to determine whether there is an association between changes in plasma lipid levels and outcomes.

Primary Outcomes:

Myocardial infarction (MI), silent MI, and CHD death.

Interventions:

Gemfibrozil (1200 mg per day) versus matching placebo.

Study Abstract:

A double-blind trial was conducted comparing gemfibrozil with placebo in 2531 men with coronary heart disease, an HDL cholesterol level of 40 mg/dL or less, and an LDL cholesterol level of 140 mg/dL or less.

The median follow-up was 5.1 years. At one year, the mean HDL was 6% higher, the mean triglyceride were 31% lower, and the mean total cholesterol was 4% lower in the gemfibrozil group than in the placebo group. LDL levels did not differ between the groups.

A primary event (MI or death) occurred in 275 of the 1267 placebo patients (21.7%) and in 219 of the 1264 gemfibrozil patients (17.3%). The overall reduction in the risk of an event was 4.4 percentage points, and the reduction in relative risk was 22% (95% confidence interval, 7% to 35%; p=0.006). A 24% relative risk reduction occurred in the combined outcome of death from coronary heart disease, nonfatal myocardial infarction, and stroke (p<0.001). Gemfibrozil therapy resulted in a significant reduction in the risk of major cardiovascular events in patients with coronary disease whose primary lipid abnormality was a low HDL cholesterol level. The findings suggest that the rate of coronary events is reduced by raising HDL cholesterol levels and lowering levels of triglycerides without lowering LDL cholesterol levels.

The major findings were published in the New England Journal of Medicine in August, 1999. A paper on lipid screening was published in the Journal of Clinical Epidemiology in July, 1999 and one on clinical implications was published in the European Heart Journal. Our cost analysis shows that gemfibrozil therapy is highly cost-effective if not cost-saving, thus providing a strong rationale for incorporating results into clinical practice. A manuscript about lipids as predictors of endpoints was published in JAMA in March, 2001. Another paper on stroke was published in Circulation in June, 2001. Dr. Robins presented data on diabetics in November, 2000 at the AHA. A paper on cost-effectiveness was published in the Archives of Internal Medicine in January 2002. A manuscript on diabetes has been accepted by the Archives of Internal Medicine.

A NHLBI grant for continuing analysis has been funded for two years. Other papers in progress include homocysteines in diabetics, fasting plasma insulin as a predictor of outcome, and the effect of lipoprotein subclass particle size on coronary events.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. male gender
2. age 73 or younger
3. presence of CHD
4. HDL-C le 40 mg/dl
5. LDL-C le 140 mg/dl
6. triglycerides le 300 mg/dl

Exclusion Criteria:

Exclusion criteria:

1. significant medical illness
2. alcohol or substance abuse
3. evidence of cholecystitis or cholelithiasis
4. ejection fraction of lt 35%
5. current use of steroids, estrogens, immunosuppressive agents, oral coagulants, or lipid modifying drug.
6. allergic to gemfibrozil or fibric acid
7. refused informed consent

Max Age: 73 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2531 (Actual)
Dates: Start 1991-06; Primary Completion 1998-09 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
incidence of nonfatal myocardial infarction or death from coronary heart disease | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hanna E. Bloomfield, MD MPH, Study Chair — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Brousseau ME, O'Connor JJ Jr, Ordovas JM, Collins D, Otvos JD, Massov T, McNamara JR, Rubins HB, Robins SJ, Schaefer EJ. Cholesteryl ester transfer protein TaqI B2B2 genotype is associated with higher HDL cholesterol levels and lower risk of coronary heart disease end points in men with HDL deficiency: Veterans Affairs HDL Cholesterol Intervention Trial. Arterioscler Thromb Vasc Biol. 2002 Jul 1;22(7):1148-54. doi: 10.1161/01.atv.0000024566.57589.2e. PMID 12117730
- [Result] Rubins HB, Robins SJ, Collins D, Fye CL, Anderson JW, Elam MB, Faas FH, Linares E, Schaefer EJ, Schectman G, Wilt TJ, Wittes J. Gemfibrozil for the secondary prevention of coronary heart disease in men with low levels of high-density lipoprotein cholesterol. Veterans Affairs High-Density Lipoprotein Cholesterol Intervention Trial Study Group. N Engl J Med. 1999 Aug 5;341(6):410-8. doi: 10.1056/NEJM199908053410604. PMID 10438259
- [Result] Rubins HB, Robins SJ, Collins D, Nelson DB, Elam MB, Schaefer EJ, Faas FH, Anderson JW. Diabetes, plasma insulin, and cardiovascular disease: subgroup analysis from the Department of Veterans Affairs high-density lipoprotein intervention trial (VA-HIT). Arch Intern Med. 2002 Dec 9-23;162(22):2597-604. doi: 10.1001/archinte.162.22.2597. PMID 12456232
- [Result] Papademetriou V, Narayan P, Rubins H, Collins D, Robins S. Influence of risk factors on peripheral and cerebrovascular disease in men with coronary artery disease, low high-density lipoprotein cholesterol levels, and desirable low-density lipoprotein cholesterol levels. HIT Investigators. Department of Veterans Affairs HDL Intervention Trial. Am Heart J. 1998 Oct;136(4 Pt 1):734-40. doi: 10.1016/s0002-8703(98)70023-7. PMID 9778079
- [Result] Rubins HB, Robins SJ, Collins D. The Veterans Affairs High-Density Lipoprotein Intervention Trial: baseline characteristics of normocholesterolemic men with coronary artery disease and low levels of high-density lipoprotein cholesterol. Veterans Affairs Cooperative Studies Program High-Density Lipoprotein Intervention Trial Study Group. Am J Cardiol. 1996 Sep 1;78(5):572-5. doi: 10.1016/s0002-9149(96)00369-4. PMID 8806347